CLINICAL TRIAL: NCT02352909
Title: A Randomised Controlled Trial on Recreational Runners With Patellofemoral Pain: Effects of Rehabilitation Approaches Based on Specific Underlying Mechanisms
Brief Title: A Controlled Trial on Recreational Runners With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-15-1 (OPPQ-REPAR); PFC-2014 (Other Grant/Funding Number: Physiotherapy Foundation of Canada, Sports Division)
Record Dates: First submitted 2014-12-03; First posted 2015-02-02 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Patellofemoral Pain (PFPS)
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Educational Status; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Education will be given on how to modify running training to encourage improvement of symptoms.
  Interventions: Other: Education
- Muscle recruitment (Experimental): Subjects will receive an additional exercise program targeting non task-specific strengthening and motor control exercises of the lower limb.
  Interventions: Other: Education; Other: Exercise program
- Reduction of knee loading (Experimental): Subjects will receive additional personalized advice on how to modify running gait in order to reduce mechanical loads at the knee (gait retraining).
  Interventions: Other: Education; Other: Gait retraining

INTERVENTIONS:
Other: Education — Education on running training modifications depending on symptoms (decrease running speed, spread running volume throughout the week, run/walk intervals, avoid downhill and stairs running). Education about symptoms will also be provided.
Other: Exercise program — A home-based program including strengthening and motor control exercises will be prescribed. The program will include 4 different phases of 2 weeks.
  Arms: Muscle recruitment
Other: Gait retraining — Running gait will be modified to reduce knee loading while running (step frequency, impact, foot strike pattern).
  Arms: Reduction of knee loading

SUMMARY:
From a rehabilitation point of view, while several approaches exist to retrain runners with PFPS, it is not clear which one is most effective, or why. The goals of this randomised-controlled trial are: 1) to compare the effectiveness of three rehabilitation programs on pain and functional limitations of runners with PFPS and 2) to explain why the programs are effective or not based on laboratory analyses. After baseline evaluation, runners will be randomly assigned to one of three treatment groups, each with a specific 8-week rehabilitation program aimed at addressing the efficiency of a specific type of retraining. These groups are: 1) Control; 2) muscle recruitment; 3) reducing knee loading during running.

The investigators hypothesis is that the intervention targeting a reduction in knee loading will be significantly more effective in reducing symptoms and improving function of runners with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Hypothesis will be tested using symptoms and functional status questionnaires. In addition, mechanistic analyses will be conducted using a running assessment using an instrumented treadmill and kinematics analyses.

ELIGIBILITY:
Inclusion Criteria:

* Running mileage at least 15km
* Symptoms since at least 3 months
* Pain level at least 3/10 during running and 3 activities among: kneeling, squatting, stairs and resisted knee extension
* Score lower than 85/100 on the KOS-ADLS

Exclusion Criteria:

* History of knee surgery or patellar dislocation
* Pain believed to originate either from meniscus or from patellar tendon
* Pain following an acute trauma
* Concurrent lower limb injuries
* History of neurological, inflammatory, rheumatoid disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms and function using a self-reported questionnaire, the Activities of Daily Living Scale of the Knee Outcome Survey (KOS-ADLS) | After 4 weeks and 8 weeks of rehabilitation; 3 months after the end of the rehabilitation program
  A validated self-reported questionnaire (found to have the best psychometric properties in this population by a systematic review; Esculier et al., Disabil Rehabil 2013;35(26):2181-90) will be used to assess the severity of symptoms and functional limitations during the activities of daily living because of knee impairment. Changes in scores to this questionnaire will allow to compare the efficacy of rehabilitation protocols.

SECONDARY OUTCOMES:
Changes in pain scores using Visual analog scales (VAS) | After 4 weeks and 8 weeks of rehabilitation; 3 months after the end of the rehabilitation program
  Visual analog scales will be used to assess levels of usual pain, worst pain and pain during running. Changes in scores to these scales will allow to compare the efficacy of rehabilitation protocols. These pain scales have been validated in this population.
Global rating of change (GRC) | After the intervention (8 weeks)
  Self-reported outcome used to monitor perception of improvement or worsening of the condition following the intervention.
Changes in the vertical loading rate of ground reaction forces during treadmill running | Baseline and after the intervention (8 weeks)
  Vertical ground reaction forces and vertical loading rate during running on a Bertec instrumented treadmill. The average and instantaneous rise in vertical ground reaction forces will be considered between initial contact and initial peak in vertical forces. Data will be collected during running between 8-10km/h on a Bertec instrumented treadmill.
Changes in ankle, knee, hip and pelvis kinematics during the stance phase of running | Baseline and after the intervention (8 weeks)
  Analysis of 3-dimensions motion of the lower limbs during running using VICON cameras. Peak angles and angular excursions will be assessed.
Changes in patellofemoral joint load during the stance phase of running | Baseline and after the intervention (8 weeks)
  Using inverse dynamics, patellofemoral joint load during the stance phase of running will be estimated by combining kinematics data with force plates data.
Changes in lower limb muscle strength | Baseline and after the intervention (8 weeks)
  Maximum isometric strength testing of the knee extensors and hip abductors, extensors and external rotators will be assessed using a handheld dynamometer with standard procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

REFERENCES:
- [Derived] Esculier JF, Bouyer LJ, Dubois B, Fremont P, Moore L, McFadyen B, Roy JS. Is combining gait retraining or an exercise programme with education better than education alone in treating runners with patellofemoral pain?A randomised clinical trial. Br J Sports Med. 2018 May;52(10):659-666. doi: 10.1136/bjsports-2016-096988. Epub 2017 May 5. PMID 28476901
- [Derived] Esculier JF, Bouyer LJ, Dubois B, Fremont P, Moore L, Roy JS. Effects of rehabilitation approaches for runners with patellofemoral pain: protocol of a randomised clinical trial addressing specific underlying mechanisms. BMC Musculoskelet Disord. 2016 Jan 6;17:5. doi: 10.1186/s12891-015-0859-9. PMID 26738470